CLINICAL TRIAL: NCT05785702
Title: The Effectiveness of Anti-wandering System on Early Spotting Residents in Unauthorized Areas Among People With Intellectual Disability: A Single Group Pre-post Test Study
Brief Title: Anti-wandering System for People With Intellectual Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Anti-wandering system_protocol
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Technology
Keywords: Gerontechnology; Anti-wandering system; Intellectual disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: The trial is a single group pre-post test study at Haven of Hope Ming Tak Day Activity Centre. There will be a pre-test of 4-6 weeks and trial of 12 weeks. During pre-test, the alarm of the anti-wandering system will be muted, and the response time in spotting participants in selected unauthorized areas without system alarm can be recorded. During the trial period, the alarm will be turned on, so that care staff will be alerted when participants enter unauthorized area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The anti-wandering system (Experimental): The experimental group will use the anti-wandering system 4-6-week of pre-test and 12-week of test trial.
  Interventions: Device: The anti-wandering system

INTERVENTIONS:
Device: The anti-wandering system — During the testing period, the system will promptly notify care staff if a participant enters unauthorized areas. A care staff will then go to that area and search for the participant. After the participant is found, care staff will reset the system, and then return the participant to a safe place.

SUMMARY:
The study has 6 research questions regarding the use of the anti-wandering system in day activity centre cum hostel for persons with intellectual disabilities:

Primary study questions:

1. Can the anti-wandering system reduce the time in seconds to turn off the alarm made by the system (a proxy measure of the response time of care staff)?
2. Can the anti-wandering system reduce the burden of care staff on keeping track of the residents?

   Secondary study questions:
3. How many alarms does the anti-wandering system generate?
4. How many false alarms does the anti-wandering system made as reported by staff?

   Auxiliary study questions:
5. What are the reasons for keeping or loosening restrictions on users due to the use of the anti-wandering system?
6. What are the perceived benefits and feasibility of anti-wandering system compared to conventional anti-wandering practices?

DETAILED DESCRIPTION:
Study design

The trial is a single group pre-post test study at Haven of Hope Ming Tak Day Activity Centre and Hostel and Haven of Hope Sau Mau Ping Day Activity Centre Cum Hostel. There will be a pre-test of 4 weeks and trial of 12 weeks. During pre-test, the alarm of the anti-wandering system will be muted, and the response time in spotting participants in selected unauthorized areas without system alarm can be recorded. During the trial period, the alarm will be turned on, so that care staff will be alerted when participants enter unauthorized area.

This protocol complies with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Guideline for Good Clinical Practice (ICH-GCP) and Declaration of Helsinki.

Procedures

1. Participants' selection and consent

   If it is feasible to install radio frequency identification (RFID) tags on all the clothes of all the residents in the study sites, all of them will be invited to participate in the trial. If this is not feasible, priority will be given to those who have higher risk in wandering (i.e. have a history of running off, attempting to leave authorized areas, or entering unauthorized areas).

   Participants and their family members will be notified about the utilization of the anti-wandering system and installation of the RFID tags in participants' clothes. If they do not want to participate, they can notify the care staff (Opt-out participation).

   For care staff, it will be presumed that they agree to participate in the study if they complete the anonymous questionnaire (i.e. implied consent) on that assesses the burden of care staff on keeping track of the residents. Written consent will be obtained from care staff before qualitative interview.
2. System installation

   The system installation includes installing the RFID sensors in the entrances of the kitchen, laundry room, storage room, activity room and pharmacy, inserting RFID tags (size about 4cm x 1cm x 0.3cm) in the participants' clothes, and installing related software(s) in computers in the general office. The service unit and the product supplier shall discuss the installation plan.
3. 1-month pre-test

   The objective of the pre-test period (Week 1 to Week 4) is to collect baseline data on the time it takes the care staff to spot a resident who has entered an unauthorized area. During the pre-test period, the alarm of the anti-wandering system will be muted. Existing anti-wandering measures will be maintained, including locking unauthorized areas, setting up carts or barriers at the entrance of the unauthorized areas, having staff stay in the unauthorized areas when the doors of the areas are open, and forbidding residents hanging around during certain time of the day. When care staff spots a resident in an unauthorized area, he or she will reset the anti-wandering system and then return the resident to a safe place. During the process, the system will record the response time of the care staff without system alarm. Reminders on contacting the general office staff to reset the anti-wandering system will be posted in unauthorized areas.
4. Training for care staff

   A few identical 1-hour training sessions will be provided to care staff. The supplier will instruct and demonstrate to care staff how to use the anti-wandering system. The University of Hong Kong (HKU) researcher will then explain the test flow and data collection. This training will be recorded so that care staff can re-watch it. A protocol with related operations will be provided to care staff.
5. Implementation

During the testing period, the system will promptly notify care staff if a participant enters unauthorized areas (e.g. the speaker installed at the hallway and monitor at the general office will broadcast and display the bed number of the participant and their position). A care staff will then go to that area and search for the participant. After the participant is found, care staff will contact the staff in the general office to reset the system, and then return the participant to a safe place. At the end of each shift, care staff will document any abnormal events, as determined by the care staff, during the use of the new anti-wandering system in a log book. HKU researcher will analyze the record to determine whether the alarm generated by the system is false or not. This experience will be used to revise the operation protocol.

Blinding

No blinding will be done for this single group study.

Sample size determination

The number of residents is estimated by the number of the residents residing in the study sites. The number of care staff is estimated by the number of related staff working in the study sites. It is expected that 40 residents and 20 care staff will be recruited.

Data analyses

1. Main analysis

   Independent sample t-test will be used to test the difference of the response time and the anonymous data of care staff burden (including the perceived frequency of giving residents freedom of movement, feeling guilt in restricting residents, having conflicts with residents due to restricting them, and worrying residents to enter unauthorized areas unsupervised) between pre-test (from Week 1 to Week 4) and main trial (from Week 5 to Week 16). Descriptive statistics will be used to examine whether the care staff have more time to handle other duties and whether they can better concentrate on other duties.
2. Process evaluations

   The number of alarms generated by the system, the number of false alarms reported by care staff, and the number of missing person report will be counted. False alarm rate will be calculated by dividing the number of false alarms by the total number of alarms.

   The reasons for keeping or loosening restrictions on users due to the use of the anti-wandering system will be summarised.
3. Qualitative interview

The interview content will be transcribed verbatim in Chinese for further analysis. The qualitative interview transcripts will be analyzed by using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the anti-wandering system. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of residents:

• Residents of the study sites

Inclusion criteria of care staff:

• Responsible for the operation of the anti-wandering system

Exclusion Criteria:

Exclusion criteria of residents:

• Not independently mobile (i.e. unable to walk around without care staff assistance)

Exclusion criteria of care staff:

• Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The time in seconds to turn off the alarm (a proxy measure of the response time of care staff in spotting residents in unauthorized areas) | From the start of pre-test to the end of the 12-week trial period
  The time in seconds from the alarm going off to the alarm being turned off will be recorded by anti-wandering system.
The burden of care staff on keeping track of the residents | Before the pre-test and the end of the 12-week trial period
  Care staff will complete five items indicating their burden in tracking of the participants under the anti-wandering system on a 5-point Likert scale (i.e. 1 indicating no burden and 5 indicating severe burden). The minimum and maximum values of the scale are 5 and 30 respectively, with higher score indicating care staff having burden. The contents include the perceived frequency of giving residents freedom of movement, feeling guilt in restricting residents, having conflicts with residents due to restricting them, and worrying residents to enter unauthorized areas unsupervised. At the end of the trial, they will fill in two additional questions of whether they have more time to handle other duties and whether they can better concentrate on other duties.

SECONDARY OUTCOMES:
The number of system alarms | From the start of 4-week pre-test to the end of the 12-week trial period
  The number of alarms will be recorded by the system and provided by supplier.
The number of false alarms reported by staff | From the start to the end of the 12-week trial period
  The number of false alarms will be reported by care staff and the perceived abnormal events will be documented by care staff in log book.
The reasons for keeping or loosening restrictions on users due to the use of the anti-wandering system | In the mid-term review meeting during the 12-week trial period
  The reasons for keeping or loosening restrictions on users due to the use of the anti-wandering system will be summarised in a mid-term meeting.
The feasibility of anti-wandering system | At the end of the 12-week trial period
  All related care staffs will complete six items indicating the feasibility in using the anti-wandering system on a 5-point Likert scale (i.e. 1 indicating difficult to use and 5 indicating easy to use).
Qualitative measures: The perceived benefits and feasibility of anti-wandering system compared to conventional anti-wandering practices in care staff | At the end of the 12-week trial period
  A total of 4 to 10 care staff / general officer will be interviewed. Interview contents include:
  1. How is the accuracy of the anti-wandering system?
  2. Can the system reduce staff workload and the mental burden?
  3. Do you think the system is safe?
  4. Is it easy to use the system?
  5. Is it easy to install the system or the RFID tag?
  6. Is there any consideration in installation of the RFID tag?
  7. What are the benefits in new anti-wandering system?
  8. Can it reduce the staff time in searching for residents?
  9. Can it increase the staff concentration in handling other workload?

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Haven of Hope Residential Service for the Disabled, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.